CLINICAL TRIAL: NCT03621982
Title: A Phase 1b, Open-label, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of Camidanlumab Tesirine (ADCT-301) as Monotherapy or in Combination in Patients With Selected Advanced Solid Tumors
Brief Title: Study of ADCT-301 in Patients With Selected Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Cami in combination with pembrolizumab in solid tumors showed signals of immunomodulatory activity. However, the signals were insufficiently compelling at the tested dose/schedule to justify continuation of the study.
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-301-103; 2019-003132-23 (EudraCT Number)
Record Dates: First submitted 2018-06-28; First posted 2018-08-09 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Head and Neck Cancer Squamous Cell Carcinoma; Non-small Cell Lung Cancer; Gastric Cancer; Esophageal Cancer; Pancreas Cancer; Bladder Cancer; Renal Cell Carcinoma; Melanoma; Triple-negative Breast Cancer; Ovarian Cancer; Colo-rectal Cancer; Fallopian Tube Cancer
Keywords: Camidanlumab tesirine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Renal Cell; Melanoma; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Colonic Neoplasms; Fallopian Tube Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADCT-301 Monotherapy (Experimental): In Part 1 (dose escalation) participants received escalating doses of ADCT-301 as monotherapy.
  Camidanlumab tesirine is administered as a 30-minute intravenous (IV) infusion on Day 1 of each cycle. Participants treated with camidanlumab tesirine as monotherapy, in the initial dose cohort will receive 20 μg/kg Q3W and the highest dose was 150 μg/kg Q3W.
  Interventions: Drug: ADCT-301
- ADCT-301 Combination Therapy (Experimental): In Part 1 (dose escalation) participants received escalating doses of ADCT-301 in combination with pembrolizamab as combination therapy.
  In Part 2 (dose expansion), participants received ADCT-301 in combination with pembrolizamab as combination therapy at the dose identified in Part 1 (dose escalation).
  Participants treated with camidanlumab tesirine in combination with pembrolizumab, in the initial dose cohort received 30 μg/kg Q3W of camidanlumab tesirine.
  Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the camidanlumab tesirine infusion).
  Interventions: Drug: ADCT-301; Biological: Pembrolizumab

INTERVENTIONS:
Drug: ADCT-301 — intravenous infusion
  Other Names: Camidanlumab tesirine
Biological: Pembrolizumab — intravenous infusion
  Other Names: Keytruda
  Arms: ADCT-301 Combination Therapy

SUMMARY:
This study evaluates ADCT-301 in patients with Selected Advanced Solid Tumors. Patients will participate in a Treatment Period with 3-week cycles and a Follow-up Period every 12 weeks for up to 1 year after treatment discontinuation.

DETAILED DESCRIPTION:
This is a Phase 1b, multi-center, open-label study with a dose-escalation part and a dose expansion part. The duration of the study participation for each participant was defined as the time from the date of signed written informed consent to the completion of the followup period, withdrawal of consent, loss to follow-up, or death, whichever occurs first.

The study was include a Screening Period (of up to 21 days), a Treatment Period (with cycles of 3 weeks for a Q3W dosing regimen), and a Follow-up Period (approximately every 12 week visits) for up to 1 year after treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any procedures.
2. Male or female participants aged 18 years or older.
3. Pathologic diagnosis of solid tumor malignancy that is locally advanced or metastatic at time of Screening:

   Part 1 Dose escalation camidanlumab tesirine as monotherapy:

   Selected advanced solid tumors: colorectal, head and neck, NSCLC, gastric and esophageal cancers, pancreas, bladder, renal cell carcinoma, melanoma, TNBC, and ovarian/fallopian tube cancers

   Part 1 Dose-escalation camidanlumab tesirine in combination with pembrolizumab:

   Selected advanced solid tumors: colorectal cancer, gastric-esophageal cancer, ovarian /fallopian tube cancer, pancreatic cancer, non-small cell lung cancer, and melanoma.

   Note: For colorectal cancer, gastric-esophageal cancer, ovarian/fallopian tube cancer, pancreatic cancers mismatch repair (MMR) / microsatellite stability (MSS) / microsatellite instability (MSI) status was mandatory. If MMR/MSS/MSI status was not available at signature of the informed consent, the test should be performed before Cycle 1 Day 1 (C1D1).

   Part 2 Dose expansion camidanlumab tesirine in combination with pembrolizumab:
   * Group 1: One of the indications identified in Part 1, for which at least 1 response (PR or CR) was seen.
   * Group 2: Participants with advanced solid tumors and MSI-H/dMMR status, who had received a prior regimen containing PD-1/PD-L1 inhibitors, for which the best response was CR, PR, or SD ≥4 months, and then progressed while under treatment with the PD-1/PD-L1 inhibitor-based regimen.

   Note: A maximum of 4 participants with the same indication was allowed in this basket group.
4. Participants who were refractory to or intolerant of existing therapy(ies) known to provide clinical benefit for their condition.
5. Participants with advanced/metastatic cancer, with measurable disease as determined by RECIST v1.1 or immune-related Response Criteria (irRC)/ immune-related Response Evaluation Criteria In Solid Tumors (irRECIST)/ immune-related Response Evaluation Criteria In Solid Tumors (iRECIST)/ immune-modified Response Evaluation Criteria in Solid Tumors (imRECIST) as per Investigator discretion.
6. A) For camidanlumab tesirine as monotherapy: Participant must have a site of disease amenable to biopsy and was willing to undergo fresh biopsy procedures (minimum 3 passes each) prior to first dose, according to the treating institution's guidelines.

   B) Participants included in the paired-biopsy cohort must in addition be willing to undergo fresh biopsy procedures (minimum 3 passes each) after receiving at least 1 dose of study drug.

   C) For camidanlumab tesirine in combination with pembrolizumab: Participant must either had a site of disease amenable to biopsy and must provide fresh tumor biopsy prior to C1D1, or have sufficient available archival tumor tissue (biopsied after their last disease progression, and in the situation where the participant had received no additional anti-cancer therapy between their progression and C1D1). Participants were must willing to undergo fresh biopsy procedures (minimum 3 passes each) after receiving at least 1 dose of study treatment, according to the treating institution's guidelines.
7. ECOG performance status 0-1.
8. Participant with life expectancy ≥ 3 months as per Investigator assessment.
9. Adequate organ function as defined by screening laboratory values within the following parameters:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^3/μL (off growth factors at least 72 hours).
   2. Platelet count ≥100 × 10^3/μL without transfusion in the past 10 days.
   3. Hemoglobin ≥9 g/dL (5.6 mmol/L) (prior transfusion allowed).
   4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or gamma glutamyl transferase (GGT) ≤2.5 × the upper limit of normal (ULN) if there is no liver involvement; ALT or AST ≤5 × ULN if there is liver involvement.
   5. Total bilirubin ≤1.5 × ULN (patients with known Gilbert's syndrome may have a total bilirubin up to ≤3 × ULN with direct bilirubin ≤1.5 × ULN).
   6. Blood creatinine ≤1.5 × ULN or calculated creatinine clearance ≥60 mL/min by the Cockcroft-Gault equation.
10. Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test within 7 days prior to start of study drug for women of childbearing potential (WOCBP).
11. Women of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 9.5 months after the last dose of camidanlumab tesirine or 4 months after last dose of pembrolizumab, whichever is the latest. Men with female partners who were of childbearing potential must agree to use a condom when sexually active or practice total abstinence from the time of giving informed consent until at least 6.5 months after the participant received the last dose of camidanlumab tesirine or 4 months after last dose of pembrolizumab, whichever was the latest.

Exclusion Criteria:

1. Participation in another investigational interventional study.
2. Prior therapy with a CD25 (IL-2R) antibody.
3. Known history of ≥Grade 3 hypersensitivity to a therapeutic antibody.
4. Participants with prior solid organ or allogeneic bone marrow transplant.
5. History of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, Sjögren's syndrome, autoimmune vasculitis [e.g., Wegener's granulomatosis]) (participants with vitiligo, type 1 diabetes mellitus, residual hypothyroidism, hypophysitis due to autoimmune condition only requiring hormone replacement may be enrolled).
6. History of neuropathy considered of autoimmune origin (e.g., polyradiculopathy including Guillain-Barré syndrome and myasthenia gravis) or other central nervous system (CNS) autoimmune disease (e.g., poliomyelitis, multiple sclerosis).
7. History of recent infection (within 4 weeks of C1D1) caused by a pathogen known to be associated with GBS, for example: herpes simplex virus 1/2 (HSV1, HSV2), varicella zoster virus (VZV), Epstein-Barr virus (EBV), cytomegalovirus (CMV), measles, Influenza A, Zika virus, Chikungunya virus, mycoplasma pneumonia, Campylobacter jejuni, enterovirus D68, or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

   Note: An influenza test and a pathogen-directed SARS-CoV-2 test (such as polymerase chain reaction [PCR]) were mandatory and must be negative before initiating study treatment (tests to be performed 3 days or less prior to dosing on C1D1; an additional 2 days were allowed in the event of logistical issues for receiving the results on time).
8. Known seropositive and requiring anti-viral therapy for human immunodeficiency (HIV) virus, hepatitis B virus (HBV), or hepatitis C virus (HCV). Note: Testing was not mandatory to be eligible but should be considered in participants with high risk for these infections; testing was mandatory if status was unknown.
9. History of Stevens-Johnson syndrome or toxic epidermal necrolysis.
10. Failure to recover to ≤Grade 1 (Common Terminology Criteria for Adverse Events version 4.0 [CTCAE version 4.0]) from acute nonhematologic toxicity (to ≤Grade 2 for neuropathy or alopecia), due to previous therapy, prior to screening.
11. Symptomatic CNS metastases or evidence of leptomeningeal disease (brain MRI or previously documented cerebrospinal fluid [CSF] cytology). Previously treated asymptomatic CNS metastases were permitted provided that the last treatment (systemic anticancer therapy and/or local radiotherapy) was completed ≥4 weeks prior to Day 1 except usage of low dose of steroids on a taper (i.e., up to 10 mg prednisone or equivalent on Day 1 and consecutive days were permissible if being tapered down). Participants with discrete dural metastases are eligible.
12. Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath).
13. Active diarrhea CTCAE Grade 2 or a medical condition associated with chronic diarrhea (such as irritable bowel syndrome, inflammatory bowel disease).
14. Active infection requiring systemic antibiotic therapy.
15. Active bleeding diathesis or significant anticoagulation (international normalized ratio [INR] ≥2.0).
16. Breastfeeding or pregnant.
17. Significant medical comorbidities, including uncontrolled hypertension (blood pressure [BP] ≥160 mmHg systolic and/or ≥110 mmHg diastolic repeatedly with or without anti hypertensive medication), unstable angina, congestive heart failure (greater than New York Heart Association class II), electrocardiographic evidence of acute ischemia, coronary angioplasty or myocardial infarction within 6 months prior to screening, severe uncontrolled atrial or ventricular cardiac arrhythmia, poorly controlled diabetes, active ulceration of the upper gastrointestinal (GI) tract or GI bleeding, or severe chronic pulmonary disease.
18. Major surgery, radiotherapy, chemotherapy or other anti-neoplastic therapy within 14 days prior to start of study drug (C1D1), except shorter if approved by the Sponsor. For cytotoxic agents that have major delayed toxicity, e.g., mitomycin C and nitrosoureas, 4 weeks is indicated as washout period. For participants received systemic anticancer immunotherapies (as opposed to intralesional) that lead to activation of Teffs and/or increase the Teff/Treg ratio, such as anti-PD-1 antibodies, 4 weeks were indicated as the washout period.
19. Use of any other experimental medication within 14 days prior to start of study drug (C1D1).
20. Participants requiring concomitant immunosuppressive agents or chronic treatment with corticosteroids except:

    * replacement dose steroids in the setting of adrenal insufficiency
    * topical, inhaled, nasal, and ophthalmic steroids are allowed.
21. Planned live vaccine within 30 days prior to the first dose of study treatment and during study treatment.
22. Congenital long QT syndrome, or a corrected QTcF interval of ≥ 480 ms, at screening (unless secondary to pacemaker or bundle branch block).
23. Active second primary malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's medical monitor and Investigator agree and document should not be exclusionary.
24. Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgment, made the participant inappropriate for study participation or put the participant at risk.
25. For participants treated with camidanlumab tesirine in combination with pembrolizumab: patients intolerant to checkpoint-inhibitor or with a history of the following ≥ Grade 3 immune-related adverse events: hepatitis, renal, ocular, neurologic, cardiovascular, rheumatologic, and hematologic.
26. For participants treated with camidanlumab tesirine in combination with pembrolizumab: participants with a history of non-infectious pneumonitis related to prior systemic treatment and that require treatment with steroids within the last 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Stanford Cancer Center, Palo Alto, California
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - Oregon Health and Science University, Portland, Oregon
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - The START Center for Cancer Care, San Antonio, Texas
- Belgium (2):
  - Institut Jules Bordet, Anderlecht
  - Universitair Ziekenhuis Gent, Ghent
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London, England
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 9 study centers in 3 countries, including the United States, Belgium, and the United Kingdom, from November 2018 to December 2022.
Pre-assignment Details: In part 1, participants were to receive escalating doses of camidanlumab tesirine as monotherapy or escalating doses of camidanlumab tesirine in combination with pembrolizumab, guided by a 3+3 design. The study was terminated prior to enrollment for Part 2 of the study.
Groups:
- ADCT-301 Monotherapy 20 µg/kg: Participants received 20 µg/kg ADCT-301 every 3 weeks (Q3W), intravenous (IV) infusion on Day 1 of each 21-day cycle.
- ADCT-301 Monotherapy 30 µg/kg: Participants received 30 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
- ADCT-301 Monotherapy 45 µg/kg: Participants received 45 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
- ADCT-301 Monotherapy 60 µg/kg: Participants received 60 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
- ADCT-301 Monotherapy 80 µg/kg: Participants received 80 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
- ADCT-301 Monotherapy 100 µg/kg: Participants received 100 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
- ADCT-301 Monotherapy 125 µg/kg: Participants received 125 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
- ADCT-301 Monotherapy 150 µg/kg: Participants received 150 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
- ADCT-301 Combination Therapy 20 µg/kg + Pembrolizamab (Pemb): Participants received 20 µg/kg ADCT-301 Q3W, IV and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combination Therapy 30 µg/kg + Pemb: Participants received 30 µg/kg ADCT-301 Q3W, IV and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combination Therapy 45 µg/kg + Pemb: Participants received 45 µg/kg ADCT-301 Q3W, IV and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combination Therapy 60 µg/kg + Pemb: Participants received 60 µg/kg ADCT-301 Q3W, IV and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combination Therapy 80 µg/kg + Pemb: Participants received 80 µg/kg ADCT-301 Q3W, IV and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combination Therapy 100 µg/kg + Pemb: Participants received 100 µg/kg ADCT-301 Q3W, IV and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
Period: Overall Study
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pembrolizamab (Pemb) | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Started | 3 | 5 | 5 | 5 | 8 | 7 | 8 | 3 | 1 | 4 | 10 | 9 | 4 | 6
Completed | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 5 | 4 | 8 | 5 | 8 | 3 | 1 | 4 | 10 | 9 | 4 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 2
Not completed — Investigator/Sponsor decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2
Not completed — Death | 2 | 4 | 4 | 3 | 8 | 4 | 6 | 3 | 0 | 3 | 8 | 4 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ADCT-301 Monotherapy 20 µg/kg: Participants received 20 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
- ADCT-301 Combination Therapy 20 µg/kg + Pemb: Participants received 20 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combination Therapy 30 µg/kg + Pemb: Participants received 30 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combination Therapy 45 µg/kg + Pemb: Participants received 45 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combination Therapy 60 µg/kg + Pemb: Participants received 60 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combination Therapy 80 µg/kg +Pemb: Participants received 80 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combination Therapy 100 µg/kg + Pemb: Participants received 100 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- Total: Total of all reporting groups
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg +Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb | Total
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 8 | 7 | 8 | 3 | 1 | 4 | 10 | 9 | 4 | 6 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4 | 3 | 4 | 2 | 6 | 3 | 0 | 3 | 5 | 2 | 2 | 4 | 42
  >=65 years | 1 | 3 | 1 | 2 | 4 | 5 | 2 | 0 | 1 | 1 | 5 | 7 | 2 | 2 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 3 | 3 | 3 | 2 | 1 | 0 | 3 | 7 | 7 | 3 | 3 | 41
  Male | 1 | 3 | 3 | 2 | 5 | 4 | 6 | 2 | 1 | 1 | 3 | 2 | 1 | 3 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 2 | 4 | 5 | 5 | 8 | 7 | 8 | 3 | 0 | 4 | 10 | 9 | 4 | 5 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  White | 3 | 4 | 4 | 4 | 7 | 7 | 8 | 3 | 0 | 4 | 7 | 9 | 3 | 5 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an AE that occurs or worsens in the period extending from the first dose of study drug to 30 days after the last dose of study drug in this study or start of a new anticancer therapy, whichever is earlier.
  Any clinically significant changes from baseline in the safety laboratory values, vital signs, 12-lead electrocardiogram (ECG), and Eastern Cooperative Oncology Group (ECOG) performance status were reported as TEAEs.
Time Frame: Up to 3 years
Population: Safety Analysis Set: The Safety analysis set consists of all participants who received study drug.
Measure: Count of Participants; unit: Participants
Groups:
- ADCT-301 Combination Therapy 80 µg/kg + Pemb; ADCT-301 Combination Therapy 100 µg/kg + Pemb: Participants received 20 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 8 | 7 | 8 | 3 | 1 | 4 | 10 | 9 | 4 | 6
Participants | 3 | 5 | 5 | 5 | 8 | 7 | 8 | 3 | 1 | 4 | 10 | 9 | 4 | 6

2. Primary Outcome: Number of Participants Who Experienced TEAEs by Common Terminology Criteria for Adverse Events (CTCAE) Grade
Description: AEs were graded according to CTCAE v4.0 (or more recent). For events not included in the CTCAE criteria, the severity of the AE was graded on a scale of 1 to 5, where 1 is asymptomatic or mild symptoms, 2 is moderate, 3 is severe, 4 is Life-threatening consequences and 5 is death related to an AE.
Time Frame: Up to 3 years
Population: Safety Analysis Set: The Safety analysis set consists of all participants who received study drug and experienced TEAEs only.
Measure: Count of Participants; unit: Participants
Groups:
- ADCT-301 Combination Therapy 80 µg/kg + Pemb: Participants received 80 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 8 | 7 | 8 | 3 | 1 | 4 | 10 | 9 | 4 | 6
Participants
  Grade 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 2 | 1
  Grade 3 | 3 | 4 | 3 | 2 | 5 | 2 | 4 | 1 | 1 | 2 | 7 | 6 | 2 | 5
  Grade 4 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 5 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Serious Adverse Events (SAEs)
Description: A SAE is defined as any AE that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization for elective procedures or for protocol compliance is not considered an SAE), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or important medical events that do not meet the preceding criteria but based on appropriate medical judgement may jeopardize the participant or may require medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: Up to 3 years
Population: Safety Analysis Set: The Safety analysis set consists of all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 8 | 7 | 8 | 3 | 1 | 4 | 10 | 9 | 4 | 6
Participants | 2 | 1 | 2 | 3 | 3 | 1 | 3 | 3 | 1 | 3 | 5 | 8 | 2 | 5

4. Primary Outcome: Number of Participants Who Experienced a SAE by CTCAE Grade
Description: AEs were graded according to CTCAE v4.0 (or more recent). For events not included in the CTCAE criteria, the severity of the AE was graded on a scale of 1 is mild or asymptomatic, 2 is moderate, 3 is severe, 4 is Life-threatening and 5 is death related to an AE.
Time Frame: Up to 3 years
Population: Safety Analysis Set: The Safety analysis set consists of all participants who received study drug. Analysis only included participants with SAEs.
Measure: Count of Participants; unit: Participants
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 2 | 1 | 2 | 3 | 3 | 1 | 3 | 3 | 1 | 3 | 5 | 8 | 2 | 5
Participants
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 | 2 | 1 | 1 | 2 | 2 | 0 | 2 | 1 | 1 | 2 | 5 | 7 | 1 | 4
  Grade 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Who Experienced a Dose Interruption
Description: Dose interruption for participants treated with ADCT-301 as monotherapy and for participants treated with ADCT-301 in combination with pembrolizumab.
Time Frame: Up to 3 years
Population: Safety Analysis Set: The Safety analysis set consists of all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 8 | 7 | 8 | 3 | 1 | 4 | 10 | 9 | 4 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants Who Experienced a Dose Reduction
Description: Dose reductions for participants treated with ADCT-301 as monotherapy and for participants treated with ADCT-301 in combination with pembrolizumab.
Time Frame: Up to 3 years
Population: Safety Analysis Set: The Safety analysis set consists of all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 8 | 7 | 8 | 3 | 1 | 4 | 10 | 9 | 4 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Description: For the dose-escalation of ADCT-301 as monotherapy, DLT is defined as any of the following events like hematologic DLT and non-hematologic DLT which occur during the 21 days following the first study drug administration period of Part 1, except those that are clearly due to underlying disease or extraneous causes.
  For the dose-escalation of ADCT-301 in combination with pembrolizumab, a DLT is defined as any of the following events ike hematologic DLT and non-hematologic DLT which occur during the 21 days following the first study drug administration period of Part 1, except those that are clearly due to underlying disease or extraneous causes.
Time Frame: Day 1 to Day 21
Population: DLT Analysis Set: The DLT-evaluable analysis set consisted of participants in Part 1 who received study drug.
Measure: Count of Participants; unit: Participants
Groups:
- ADCT-301 Combined Therapy 20 µg/kg + Pemb: Participants received 20 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combined Therapy 30 µg/kg + Pemb: Participants received 30 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combined Therapy 45 µg/kg + Pemb: Participants received 45 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combined Therapy 60 µg/kg + Pemb: Participants received 60 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combined Therapy 80 µg/kg + Pemb: Participants received 80 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
- ADCT-301 Combined Therapy 100 µg/kg + Pemb: Participants received 100 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combined Therapy 20 µg/kg + Pemb | ADCT-301 Combined Therapy 30 µg/kg + Pemb | ADCT-301 Combined Therapy 45 µg/kg + Pemb | ADCT-301 Combined Therapy 60 µg/kg + Pemb | ADCT-301 Combined Therapy 80 µg/kg + Pemb | ADCT-301 Combined Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 8 | 7 | 8 | 3 | 1 | 4 | 10 | 9 | 4 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1

8. Secondary Outcome: Overall Response Rate (ORR) According to the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Description: The ORR was defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). The overall response category was derived based on response assessment performed on or before the start of subsequent anti-cancer therapy.
Time Frame: Up to 3 years
Population: Efficacy Analysis Set: The Efficacy analysis set consisted of all participants who received at least 1 dose of study drug, had valid Baseline disease assessment(s), and at least one valid post-Baseline disease assessment. Participants who did not have a post-Baseline assessment due to early clinical progression or death (after receiving study drug) were also included. The monotherapy arms and combination arms were pooled as pre-specified in protocol section 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ADCT-301 Monotherapy: Participants received 20, 30, 45, 60, 80, 100, 125 and 150 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
- ADCT-301 Combination Therapy: Participants received 20, 30, 45, 60, 80 and 100 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
Arm/Group | ADCT-301 Monotherapy | ADCT-301 Combination Therapy
Number analyzed (Participants) | 44 | 33
percentage of participants | 0 [0 to 0] | 15.2 [5.1 to 31.9]

9. Secondary Outcome: Duration of Response (DOR) as Per RECIST v 1.1
Description: DOR is defined among objective responders (CR or PR) as the time from the earliest date of first response until the first date of either disease progression (based on radiographic or clinical progression at end of treatment [EOT]/end of study [EOS]) or death due to any cause.
Time Frame: Up to 3 years
Population: Efficacy Analysis Set: This analysis set consisted of all participants who received at least 1 dose of study drug, had valid Baseline disease assessment(s), and at least one valid post-Baseline disease assessment. Participants who did not have a post-Baseline assessment due to early clinical progression or death were also included. The monotherapy arms and combination arms were pooled as pre-specified in protocol section 3.
  Includes participants who experienced CR or PR only.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- ADCT-301 Combination Therapy: Participants received 20, 30, 45, 60, 80, 100 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
Arm/Group | ADCT-301 Monotherapy | ADCT-301 Combination Therapy
Number analyzed (Participants) | 0 | 5
months |  | 9.26 [3.15 to NA] — Upper limit could not be calculated as not enough participants achieved a response.

10. Secondary Outcome: Progression-free Survival (PFS) as Per RECIST v 1.1
Description: PFS defined as the time between start of treatment and the first documentation of recurrence, progression, or death for participants treated with ADCT-301 as monotherapy and for participants treated with ADCT-301 in combination with pembrolizumab.
Time Frame: Up to 3 years
Population: Efficacy Analysis Set: The Efficacy analysis set consisted of all participants who received at least 1 dose of study drug, had valid Baseline disease assessment(s), and at least one valid post-Baseline disease. The monotherapy arms and combination arms were pooled as pre-specified in protocol section 3.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- ADCT-301 Monotherapy: Participants received 20,30, 45, 60, 100, 125 and 150 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
- ADCT-301 Combination Therapy: Participants received 20, 30, 45, 60,80,100,125 and 150 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
Arm/Group | ADCT-301 Monotherapy | ADCT-301 Combination Therapy
Number analyzed (Participants) | 44 | 33
months | 1.35 [1.18 to 1.38] | 1.41 [1.25 to 2.10]

11. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time between the start of treatment and death from any cause for participants treated with ADCT-301 as monotherapy and for participants treated with ADCT-301 in combination with pembrolizumab.
Time Frame: Up to 3 years
Population: Efficacy Analysis Set: The Efficacy analysis set consisted of all participants who received at least 1 dose of study drug, had valid Baseline disease assessment(s), and at least one valid post-Baseline disease assessment. The monotherapy arms and combination arms were pooled as pre-specified in protocol section 3.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- ADCT-301 Combination Therapy: Participants received 20, 30, 45, 60, 80, 100, 125 and 150 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
Arm/Group | ADCT-301 Monotherapy | ADCT-301 Combination Therapy
Number analyzed (Participants) | 44 | 33
months | 4.37 [2.99 to 6.74] | 7.59 [4.11 to 10.61]

12. Secondary Outcome: Time to Maximum Concentration (Tmax) of ADCT-301 in Serum Total Antibody, PBD-conjugated Antibody, and Unconjugated Warhead SG3199
Description: The pharmacokinetic (PK) profile included determination of Tmax in serum Total antibody, PBD-conjugated antibody, and unconjugated warhead SG3199. For participants treated with camidanlumab tesirine in combination with pembrolizumab, the collection of PK data was stopped upon consultation with the Sponsor if ADCT-301 administration is discontinued and pembrolizumab continues.
  Upon consultation with the Sponsor, no further PK samples were collected, ADCT-301 was permanently discontinued and pembrolizumab continues as single agent.
Time Frame: Cycle 1 Day 1 (C1D1), from Pre-dose to 4 hr, 96 hr, 168 hr and 336 hr post dose; Cycle 2 Day 1 (C2D1), from Pre-dose to 4 hr, 48 hr, 96 hr, 168 hr and 336 hr post dose
Population: PK Analysis Set: The PK analysis set consisted of all participants who received study drug and had at least 1 pre-C1D1 and 1 post-dose valid assessment. Includes participants with available data at each timepoint.
  The overall number of participants analyzed represents the number of participants with available PK data at any timepoint.
  Includes participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 8 | 7 | 7 | 3 | 1 | 4 | 10 | 9 | 4 | 6
days
  Conjugated Antibody Cycle 1 | 0.0750 (81.1) | 0.0770 (82.4) | 0.0780 (76.2) | 0.0940 (54.8) | 0.0560 (50.3) | 0.0760 (37.0) | 0.0840 (48.6) | 0.0770 (87.8) | 0.0350 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.0290 (15.9) | 0.0720 (1522) | 0.108 (114) | 0.0620 (163) | 0.121 (90.2)
  Total Antibody Cycle 1 | 0.0750 (81.1) | 0.0980 (87.2) | 0.0780 (76.2) | 0.0730 (54.2) | 0.0790 (70.2) | 0.0910 (56.3) | 0.0700 (43.1) | 0.121 (65.9) | 0.0350 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.0430 (112) | 0.0830 (112) | 0.112 (99.6) | 0.0620 (163) | 0.121 (90.2)
  Unconjugated SG3199 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 6 | 1 | 0 | 0 | 1 | 1 | 2 | 3
  Unconjugated SG3199 Cycle 1 |  |  |  |  | 0.146 (37.8) | 0.116 (54.4) | 0.192 (18.6) | 0.160 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. |  |  | 2.84 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.178 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.161 (1.52) | 0.0890 (152)
  Conjugated Antibody Cycle 2: number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 5 | 4 | 3 | 1 | 3 | 7 | 7 | 3 | 3
  Conjugated Antibody Cycle 2 | 0.0670 (193) | 0.0280 (33.1) | 0.0720 (130) | 0.115 (94.2) | 0.0280 (15.7) | 0.0540 (78.3) | 0.0310 (1.12) | 0.0470 (160) | 0.0330 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.0740 (92.5) | 0.110 (542) | 0.0590 (131) | 0.0510 (147) | 0.171 (9.93)
  Total Antibody Cycle 2: number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 5 | 4 | 3 | 1 | 3 | 7 | 7 | 3 | 3
  Total Antibody Cycle 2 | 0.0670 (193) | 0.0280 (33.1) | 0.0440 (122) | 0.0760 (115) | 0.112 (91.9) | 0.0550 (79.5) | 0.0310 (1.12) | 0.0860 (173) | 0.0330 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.0740 (92.5) | 0.0690 (112) | 0.102 (106) | 0.101 (130) | 0.171 (9.93)
  Unconjugated SG3199 Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 1
  Unconjugated SG3199 Cycle 2 |  |  |  | 0.168 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.174 (0) | 0.280 (4298) | 0.170 (3.17) |  |  |  | 1.12 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.169 (2.32) | 0.0320 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.161 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation.

13. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) of ADCT-301 in Serum Total Antibody, PBD-conjugated Antibody, and Unconjugated Warhead SG3199
Description: PK profile included AUC0-last of ADCT-301 in Serum total antibody, PBD-conjugated antibody, and unconjugated warhead SG3199. For participants treated with ADCT-301 in combination with pembrolizumab, the collection of PK data was stopped upon consultation with the Sponsor if ADCT-301 administration was discontinued and pembrolizumab continues.
  Upon consultation with the Sponsor, no further PK samples were collected, ADCT-301 was permanently discontinued and pembrolizumab continues as single agent.
Time Frame: C1D1, from Pre-dose to 4 hr, 96 hr, 168 hr and 336 hr post dose; C2D1, from Pre-dose to 4 hr, 48 hr, 96 hr, 168 hr and 336 hr post dose
Population: PK Analysis Set: The PK analysis set consisted of all participants who received study drug and had at least 1 pre-C1D1 and 1 post-dose valid assessment.
  The overall number of participants analyzed represents the number of participants with available PK data at any timepoint.
  Includes participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 8 | 7 | 7 | 3 | 1 | 4 | 10 | 9 | 4 | 6
day*ng/mL
  Conjugated Antibody Cycle 1 | 229 (520) | 464 (65.8) | 484 (224) | 2067 (93.6) | 1954 (31.9) | 3440 (66.6) | 5848 (53.5) | 5571 (61.9) | 564 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 655 (53.6) | 1124 (47.0) | 1737 (35.6) | 814 (428) | 3863 (33.3)
  Total Antibody Cycle 1 | 294 (598) | 636 (113) | 647 (222) | 2857 (67.7) | 3025 (37.0) | 4938 (67.4) | 8812 (74.6) | 9078 (48.4) | 955 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 965 (73.7) | 1508 (52.7) | 2470 (42.1) | 1172 (557) | 7274 (24.0)
  Unconjugated SG3199 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 6 | 1 | 0 | 0 | 1 | 1 | 2 | 3
  Unconjugated SG3199 Cycle 1 |  |  |  |  | 0.00100 (322) | 0.00600 (751) | 0.00300 (298) | 0.00100 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. |  |  | 0.0110 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.00100 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.00100 (57.2) | 0.00200 (228)
  Conjugated Antibody Cycle 2: number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 5 | 4 | 3 | 1 | 3 | 7 | 7 | 3 | 3
  Conjugated Antibody Cycle 2 | 588 (17.3) | 676 (92.4) | 898 (95.5) | 2386 (126) | 2668 (44.0) | 4025 (101) | 8305 (22.0) | 6599 (46.1) | 2421 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 825 (37.6) | 1392 (57.0) | 1716 (84.6) | 1386 (145) | 4535 (66.2)
  Total Antibody Cycle 2: number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 5 | 4 | 3 | 1 | 3 | 7 | 7 | 3 | 3
  Total Antibody Cycle 2 | 769 (14.6) | 880 (107) | 1060 (105) | 3740 (116) | 4910 (35.8) | 5815 (72.2) | 11879 (18.8) | 9027 (48.0) | 4796 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1128 (47.5) | 1653 (57.3) | 2609 (74.9) | 3203 (41.3) | 7077 (44.1)
  Unconjugated SG3199 Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 1
  Unconjugated SG3199 Cycle 2 |  |  |  | 0.00100 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.00400 (1630) | 0.00200 (14068) | 0.0320 (3.13) |  |  |  | 0.00600 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.00300 (293) | 0.00300 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.00100 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation.

14. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) of ADCT-301 in Serum Total Antibody, PBD-conjugated Antibody, and Unconjugated Warhead SG3199
Description: The PK profile included AUCinf of ADCT-301 in serum total antibody, PBD-conjugated antibody, and unconjugated warhead SG3199. For participants treated with ADCT-301 in combination with pembrolizumab, the collection of PK data was stopped upon consultation with the Sponsor if ADCT-301 administration was discontinued and pembrolizumab continues.
  Upon consultation with the Sponsor, no further PK samples were collected, ADCT-301 was permanently discontinued and pembrolizumab continues as single agent.
Time Frame: C1D1, from Pre-dose to 4hr, 96hr, 168 hr and 336 hr post dose; C2D1, from Pre-dose to 4 hr, 48 hr, 96 hr, 168 hr and 336 hr post dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/L
Groups:
- ADCT Combination Therapy 45 µg/kg + Pemb: Participants received 45 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle and Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion).
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 1 | 2 | 2 | 4 | 7 | 7 | 6 | 3 | 1 | 1 | 4 | 8 | 2 | 6
day*µg/L
  Conjugated Antibody Cycle 1: number analyzed (Participants) | 1 | 2 | 2 | 4 | 7 | 7 | 6 | 2 | 1 | 1 | 3 | 8 | 2 | 6
  Conjugated Antibody Cycle 1 | 823 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 907 (26.6) | 1000 (14.7) | 2552 (98.1) | 2259 (30.1) | 3708 (66.0) | 7420 (30.9) | 8031 (22.6) | 678 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 873 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 2058 (19.7) | 2059 (30.1) | 2725 (51.5) | 4556 (34.4)
  Total Antibody Cycle 1: number analyzed (Participants) | 1 | 0 | 2 | 2 | 6 | 5 | 5 | 3 | 0 | 1 | 4 | 5 | 2 | 3
  Total Antibody Cycle 1 | 1068 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. |  | 1331 (2.40) | 5768 (10.7) | 3962 (21.8) | 6594 (36.2) | 13018 (40.3) | 9578 (50.1) |  | 2107 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 2083 (18.4) | 3552 (23.6) | 4157 (77.3) | 7077 (8.27)
  Unconjugated SG3199 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Conjugated Antibody Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Antibody Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unconjugated SG3199 Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the End of the Dosing Interval (AUCtau) ADCT-301 in Serum Total Antibody, PBD-conjugated Antibody, and Unconjugated Warhead SG3199
Description: The PK profile included AUCtau ADCT-301 in serum total antibody, PBD-conjugated antibody, and unconjugated warhead SG3199. For participants treated with ADCT-301 in combination with pembrolizumab, the collection of PK data was stopped upon consultation with the Sponsor if ADCT-301 administration was discontinued and pembrolizumab continues.
  Upon consultation with the Sponsor, no further PK samples were collected, ADCT-301 was permanently discontinued and pembrolizumab continues as single agent.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/L
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 1 | 4 | 2 | 4 | 4 | 5 | 4 | 3 | 1 | 2 | 5 | 6 | 2 | 3
day*µg/L
  Conjugated Antibody Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total Antibody Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unconjugated SG3199 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Conjugated Antibody Cycle 2: number analyzed (Participants) | 1 | 4 | 1 | 3 | 4 | 4 | 4 | 3 | 1 | 2 | 4 | 6 | 2 | 3
  Conjugated Antibody Cycle 2 | 1776 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1110 (70.5) | 1516 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 3719 (132) | 2956 (47.2) | 6084 (26.4) | 9238 (27.5) | 7885 (31.4) | 2882 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1171 (5.95) | 1816 (46.1) | 2467 (44.6) | 2975 (18.4) | 5440 (64.1)
  Total Antibody Cycle 2: number analyzed (Participants) | 1 | 4 | 2 | 4 | 4 | 5 | 4 | 2 | 1 | 2 | 5 | 5 | 2 | 3
  Total Antibody Cycle 2 | 2562 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1302 (88.4) | 2217 (34.2) | 4490 (110) | 5565 (35.4) | 6486 (80.0) | 13483 (22.9) | 12197 (40.7) | 5399 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1856 (4.69) | 2861 (43.3) | 3720 (47.5) | 4887 (27.6) | 8920 (45.4)
  Unconjugated SG3199 Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Accumulation Index (AI) of ADCT-301 in Serum Total Antibody, PBD-conjugated Antibody and Unconjugated Warhead SG3199
Description: The PK profile included AI of ADCT-301 in serum total antibody and PBD-conjugated antibody. For participants treated with ADCT-301 in combination with pembrolizumab, the collection of PK data was stopped upon consultation with the Sponsor if ADCT-301 administration was discontinued and pembrolizumab continues.
  AI is the ratio of accumulation of a drug under steady state conditions (i.e., after repeated administration) as compared to a single dose.
  Upon consultation with the Sponsor, no further PK samples were collected, ADCT-301 was permanently discontinued and pembrolizumab continues as single agent.
Time Frame: C2D1, from Pre-dose to 4 hr, 48 hr, 96 hr, 168 hr and 336 hr post dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 1 | 3 | 2 | 4 | 4 | 5 | 4 | 3 | 1 | 2 | 5 | 6 | 2 | 3
ratio
  Conjugated Antibody Cycle 2: number analyzed (Participants) | 1 | 3 | 1 | 3 | 4 | 4 | 4 | 3 | 1 | 2 | 4 | 6 | 2 | 3
  Conjugated Antibody Cycle 2 | 1.00 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.00 (0.175) | 1.00 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.09 (7.42) | 1.01 (0.621) | 1.02 (2.41) | 1.04 (4.67) | 1.03 (2.39) | 1.00 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.00 (0.123) | 1.01 (1.05) | 1.00 (0.570) | 1.00 (0.258) | 1.02 (1.28)
  Total Antibody Cycle 2: number analyzed (Participants) | 1 | 3 | 2 | 4 | 4 | 5 | 4 | 2 | 1 | 2 | 5 | 5 | 2 | 3
  Total Antibody Cycle 2 | 1.00 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.00 (0.248) | 1.00 (0.124) | 1.03 (3.59) | 1.01 (0.819) | 1.02 (3.12) | 1.05 (6.87) | 1.05 (4.03) | 1.10 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.00 (0.257) | 1.03 (3.73) | 1.00 (0.305) | 1.01 (0.757) | 1.04 (3.01)
  Unconjugated SG3199 Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Clearance (CL) of ADCT-301 in Serum Total Antibody, PBD-conjugated Antibody and Unconjugated Warhead SG3199
Description: The PK profile included the CL of ADCT-301 in serum total antibody and PBD-conjugated antibody. For participants treated with ADCT-301 in combination with pembrolizumab, the collection of PK data was stopped upon consultation with the Sponsor if ADCT-301 administration was discontinued and pembrolizumab continues.
  Upon consultation with the Sponsor, no further PK samples were collected, ADCT-301 was permanently discontinued and pembrolizumab continues as single agent.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 1 | 4 | 2 | 4 | 7 | 7 | 6 | 3 | 1 | 2 | 5 | 8 | 2 | 6
L/day
  Conjugated Antibody Cycle 1: number analyzed (Participants) | 1 | 2 | 2 | 4 | 7 | 7 | 6 | 2 | 1 | 1 | 3 | 8 | 2 | 6
  Conjugated Antibody Cycle 1 | 0.940 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.85 (74.0) | 2.92 (15.9) | 1.37 (60.5) | 2.04 (18.3) | 1.84 (52.7) | 1.22 (16.4) | 1.36 (12.8) | 2.53 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 2.30 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.35 (22.6) | 1.33 (34.4) | 1.46 (40.3) | 1.36 (31.5)
  Total Antibody Cycle 1: number analyzed (Participants) | 1 | 0 | 2 | 2 | 6 | 5 | 5 | 3 | 0 | 1 | 4 | 5 | 2 | 3
  Total Antibody Cycle 1 | 0.869 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. |  | 2.60 (3.98) | 0.928 (0.345) | 1.35 (27.8) | 1.24 (32.8) | 0.880 (27.4) | 1.16 (18.9) |  | 1.15 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.27 (21.0) | 1.12 (24.4) | 1.14 (63.2) | 0.809 (13.1)
  Conjugated Antibody Cycle 2: number analyzed (Participants) | 1 | 4 | 1 | 3 | 4 | 4 | 4 | 3 | 1 | 2 | 4 | 6 | 2 | 3
  Conjugated Antibody Cycle 2 | 0.544 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 2.02 (69.3) | 1.91 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.01 (105) | 1.57 (18.3) | 1.18 (21.2) | 1.02 (19.9) | 1.16 (17.3) | 1.82 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 2.11 (6.07) | 1.44 (35.4) | 1.43 (43.1) | 1.47 (10.9) | 1.23 (30.7)
  Total Antibody Cycle 2: number analyzed (Participants) | 1 | 4 | 2 | 4 | 4 | 5 | 4 | 2 | 1 | 2 | 5 | 5 | 2 | 3
  Total Antibody Cycle 2 | 0.449 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 2.05 (86.9) | 1.43 (48.0) | 1.02 (88.1) | 0.994 (20.9) | 1.25 (64.9) | 0.830 (15.4) | 1.04 (26.5) | 1.16 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.58 (16.8) | 1.08 (28.9) | 1.13 (36.7) | 1.07 (19.8) | 0.890 (15.3)
  Unconjugated SG3199 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unconjugated SG3199 Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Apparent Terminal Elimination Half-life (Thalf) of ADCT-301 in Serum Total Antibody, PBD-conjugated Antibody, and Unconjugated Warhead SG3199
Description: The PK profile included the Thalf of ADCT-301 in serum total antibody and PBD-conjugated antibody. For participants treated with ADCT-301 in combination with pembrolizumab, the collection of PK data was stopped upon consultation with the Sponsor if ADCT-301 administration was discontinued and pembrolizumab continues.
  Upon consultation with the Sponsor, no further PK samples were collected, ADCT-301 was permanently discontinued and pembrolizumab continues as single agent.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 1 | 3 | 2 | 4 | 7 | 7 | 6 | 3 | 1 | 2 | 5 | 8 | 2 | 6
days
  Conjugated Antibody Cycle 1: number analyzed (Participants) | 1 | 2 | 2 | 4 | 7 | 7 | 6 | 2 | 1 | 1 | 3 | 8 | 2 | 6
  Conjugated Antibody Cycle 1 | 1.39 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.93 (40.1) | 1.49 (5.47) | 2.41 (75.5) | 1.96 (9.91) | 2.30 (54.5) | 3.66 (44.5) | 3.97 (17.9) | 1.55 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.42 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 2.64 (12.8) | 1.93 (20.8) | 2.61 (9.30) | 2.89 (41.8)
  Total Antibody Cycle 1: number analyzed (Participants) | 1 | 0 | 2 | 2 | 6 | 5 | 5 | 3 | 0 | 1 | 4 | 5 | 2 | 3
  Total Antibody Cycle 1 | 1.41 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. |  | 1.36 (11.2) | 3.22 (22.8) | 1.95 (13.7) | 2.49 (43.2) | 3.78 (42.4) | 2.79 (70.8) |  | 2.33 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 2.16 (16.8) | 2.10 (20.0) | 2.55 (13.0) | 3.00 (18.9)
  Conjugated Antibody Cycle 2: number analyzed (Participants) | 1 | 3 | 1 | 3 | 4 | 4 | 4 | 3 | 1 | 2 | 4 | 6 | 2 | 3
  Conjugated Antibody Cycle 2 | 1.75 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.89 (25.6) | 1.88 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 3.95 (118) | 2.49 (29.0) | 3.15 (43.5) | 4.08 (33.4) | 3.28 (51.7) | 2.60 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.85 (31.9) | 2.54 (42.4) | 2.24 (29.7) | 2.30 (21.4) | 3.32 (20.0)
  Total Antibody Cycle 2: number analyzed (Participants) | 1 | 3 | 2 | 4 | 4 | 5 | 4 | 2 | 1 | 2 | 5 | 5 | 2 | 3
  Total Antibody Cycle 2 | 2.22 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 1.99 (27.1) | 2.10 (17.4) | 2.86 (66.3) | 2.67 (29.1) | 2.58 (79.1) | 3.92 (48.2) | 4.70 (27.6) | 6.09 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 2.37 (18.7) | 3.13 (47.0) | 2.24 (22.5) | 2.97 (20.1) | 3.98 (35.1)
  Unconjugated SG3199 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unconjugated SG3199 Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Maximum Concentration (Cmax) of ADCT-301 in Serum Total Antibody, PBD-conjugated Antibody and Unconjugated Warhead SG3199
Description: The PK profile included determination of Cmax in serum Total antibody, PBD-conjugated Antibody and Unconjugated Warhead SG3199. For participants treated with ADCT-301 in combination with pembrolizumab, the collection of PK data was stopped upon consultation with the Sponsor if ADCT-301 administration was discontinued and pembrolizumab continues.
  Upon consultation with the Sponsor, no further PK samples were collected, ADCT-301 was permanently discontinued and pembrolizumab continues as single agent.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT-301 Combination Therapy 45 µg/kg + Pemb | ADCT-301 Combination Therapy 60 µg/kg + Pemb | ADCT-301 Combination Therapy 80 µg/kg + Pemb | ADCT-301 Combination Therapy 100 µg/kg + Pemb
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 8 | 7 | 7 | 3 | 1 | 4 | 10 | 9 | 4 | 6
µg/L
  Conjugated Antibody Cycle 1 | 317 (33.2) | 314 (34.2) | 433 (35.0) | 889 (34.3) | 901 (33.6) | 1328 (38.0) | 2017 (20.4) | 1990 (1.73) | 408 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 389 (31.3) | 594 (46.2) | 750 (17.1) | 954 (75.0) | 1937 (150)
  Total Antibody Cycle 1 | 411 (39.2) | 377 (35.7) | 552 (31.5) | 1077 (23.7) | 1270 (28.6) | 1740 (32.5) | 2442 (25.6) | 2228 (18.2) | 488 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 507 (25.8) | 719 (39.2) | 946 (18.8) | 1209 (76.2) | 2836 (126)
  Unconjugated SG3199 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 6 | 1 | 0 | 0 | 1 | 1 | 2 | 3
  Unconjugated SG3199 Cycle 1 |  |  |  |  | 0.0120 (28.3) | 0.0170 (35.8) | 0.0140 (21.8) | 0.0140 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. |  |  | 0.0110 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.0120 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.0130 (5.97) | 0.0250 (185)
  Conjugated Antibody Cycle 2: number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 5 | 4 | 3 | 1 | 3 | 7 | 7 | 3 | 3
  Conjugated Antibody Cycle 2 | 405 (12.8) | 448 (109) | 497 (28.6) | 999 (78.3) | 939 (34.5) | 1527 (43.7) | 2150 (11.1) | 2208 (13.2) | 1270 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 407 (43.0) | 603 (38.5) | 862 (82.7) | 1089 (125) | 1297 (46.4)
  Total Antibody Cycle 2: number analyzed (Participants) | 2 | 5 | 4 | 4 | 4 | 5 | 4 | 3 | 1 | 3 | 7 | 7 | 3 | 3
  Total Antibody Cycle 2 | 490 (2.60) | 560 (122) | 592 (24.7) | 1420 (62.3) | 1354 (22.9) | 1797 (35.1) | 2624 (2.67) | 2907 (7.98) | 1660 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 463 (44.6) | 745 (29.7) | 1149 (71.1) | 1355 (128) | 1690 (24.9)
  Unconjugated SG3199 Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 1
  Unconjugated SG3199 Cycle 2 |  |  |  | 0.0130 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.0130 (3.82) | 0.0110 (3.23) | 0.0170 (8.29) |  |  |  | 0.0100 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.0100 (26.4) | 0.0190 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation. | 0.0120 (NA) — Data not available due to insufficient number of observations to determine geometric coefficient of variation.

20. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) Response in Serum
Description: ADA testing included number of participants with positive pre-dose ADA response, number of participants with post-dose ADA response only, and number of participants with positive ADA response at any time. Collection of ADA was stopped if ADCT-301 administration was discontinued. For participants treated with ADCT-301 in combination with pembrolizumab, unless there was a penultimate observation of positive ADA response, no other collection of ADA data was necessary if ADCT-301 administration was discontinued.
  Upon consultation with the Sponsor, ADA samples were not collected anymore if ADCT-301 was permanently discontinued and pembrolizumab continues as single agent.
Time Frame: C1D1, from Pre-dose to 336 hr post dose.
Population: Pharmacodynamic Analysis Set: The pharmacodynamic analysis set consisted of all participants who received study drug and had at least 1 valid pharmacodynamics/biomarker assessment. The data was pooled overall as pre-specified in protocol.
  Includes participants with available data at each timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: Participants received 20, 30, 45, 60, 80, 100, 125 and 150 µg/kg ADCT-301 Q3W, IV infusion on Day 1 of each 21-day cycle.
  Pembrolizumab was administered as a 30 minute IV infusion at a fixed dose of 200 mg (starting 1 hour after the end of the ADCT-301 infusion)
Arm/Group | Overall Study
Number analyzed (Participants) | 78
Participants
  Positive ADA predose | 1
  Positive ADA post dose | 0
  Positive ADA at any time | 1
  Positive ADA before and after dose | 1

ADVERSE EVENTS:
Time Frame: All SAEs and AEs were collected from the time the participant signs the ICF until 30 days after the last dose of study drug up to a maximum of 3 years.
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have to have a causal relationship with this treatment.
Groups:
- ADCT-301 Monotherapy 20 µg/kg: Part 1 (dose escalation): 20 μg/kg; Q3W; IV A treatment cycle was defined as 3 weeks (i.e., 21 days). Infusion on Day 1 of each cycle starting from Cycle 1 onwards.
- ADCT-301 Monotherapy 30 µg/kg: Part 1 (dose escalation): 30 μg/kg; Q3W; IV A treatment cycle was defined as 3 weeks (i.e., 21 days). Infusion on Day 1 of each cycle starting from Cycle 1 onwards.
- ADCT-301 Monotherapy 45 µg/kg: Part 1 (dose escalation): 45 μg/kg; Q3W; IV A treatment cycle was defined as 3 weeks (i.e., 21 days). Infusion on Day 1 of each cycle starting from Cycle 1 onwards.
- ADCT-301 Monotherapy 60 µg/kg: Part 1 (dose escalation): 60 μg/kg; Q3W; IV A treatment cycle was defined as 3 weeks (i.e., 21 days). Infusion on Day 1 of each cycle starting from Cycle 1 onwards.
- ADCT-301 Monotherapy 80 µg/kg: Part 1 (dose escalation): 80 μg/kg; Q3W; IV A treatment cycle was defined as 3 weeks (i.e., 21 days). Infusion on Day 1 of each cycle starting from Cycle 1 onwards.
- ADCT-301 Monotherapy 100 µg/kg: Part 1 (dose escalation): 100 μg/kg; Q3W; IV A treatment cycle was defined as 3 weeks (i.e., 21 days). Infusion on Day 1 of each cycle starting from Cycle 1 onwards.
- ADCT-301 Monotherapy 125 µg/kg: Part 1 (dose escalation): 125 μg/kg; Q3W; IV A treatment cycle was defined as 3 weeks (i.e., 21 days). Infusion on Day 1 of each cycle starting from Cycle 1 onwards.
- ADCT-301 Monotherapy 150 µg/kg: Part 1 (dose escalation): 150 μg/kg; Q3W; IV A treatment cycle was defined as 3 weeks (i.e., 21 days). Infusion on Day 1 of each cycle starting from Cycle 1 onwards.
- ADCT-301 Combination Therapy 20 µg/kg + Pemb: Participants received ADCT-301 in combination with pembrolizamab as combination therapy at the dose identified in Part 1 (dose escalation) 20 µg/kg.
  Pembrolizumab at dose of 200 mg Q3W; IV was administered on Day 1 of each cycle starting from Cycle 1 onwards (dosing schedule 1).
- ADCT-301 Combination Therapy 30 µg/kg + Pemb: Participants received ADCT-301 in combination with pembrolizamab as combination therapy at the dose identified in Part 1 (dose escalation) 30 µg/kg.
  Pembrolizumab at dose of 200 mg Q3W; IV was administered on Day 1 of each cycle starting from Cycle 1 onwards (dosing schedule 1).
- ADCT Combination Therapy 45 µg/kg + Pemb: Participants received ADCT-301 in combination with pembrolizamab as combination therapy at the dose identified in Part 1 (dose escalation) 45 µg/kg.
  Pembrolizumab at dose of 200 mg Q3W; IV was administered on Day 1 of each cycle starting from Cycle 1 onwards (dosing schedule 1).
- ADCT Combination Therapy 60 µg/kg + Pemb: Participants received ADCT-301 in combination with pembrolizamab as combination therapy at the dose identified in Part 1 (dose escalation) 60 µg/kg.
  Pembrolizumab at dose of 200 mg Q3W; IV was administered on Day 1 of each cycle starting from Cycle 1 onwards (dosing schedule 1).
- ADCT Combination Therapy 80 µg/kg + Pemb: Participants received ADCT-301 in combination with pembrolizamab as combination therapy at the dose identified in Part 1 (dose escalation) 80 µg/kg.
  Pembrolizumab at dose of 200 mg Q3W; IV was administered on Day 1 of each cycle starting from Cycle 1 onwards (dosing schedule 1).
- ADCT Combination Therapy 100 µg/kg + Pemb: Participants received ADCT-301 in combination with pembrolizamab as combination therapy at the dose identified in Part 1 (dose escalation) 100 µg/kg.
  Pembrolizumab at dose of 200 mg Q3W; IV was administered on Day 1 of each cycle starting from Cycle 1 onwards (dosing schedule 1).
Arm/Group | ADCT-301 Monotherapy 20 µg/kg | ADCT-301 Monotherapy 30 µg/kg | ADCT-301 Monotherapy 45 µg/kg | ADCT-301 Monotherapy 60 µg/kg | ADCT-301 Monotherapy 80 µg/kg | ADCT-301 Monotherapy 100 µg/kg | ADCT-301 Monotherapy 125 µg/kg | ADCT-301 Monotherapy 150 µg/kg | ADCT-301 Combination Therapy 20 µg/kg + Pemb | ADCT-301 Combination Therapy 30 µg/kg + Pemb | ADCT Combination Therapy 45 µg/kg + Pemb | ADCT Combination Therapy 60 µg/kg + Pemb | ADCT Combination Therapy 80 µg/kg + Pemb | ADCT Combination Therapy 100 µg/kg + Pemb
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/5 | 4/5 | 3/5 | 8/8 | 4/7 | 6/8 | 3/3 | 0/1 | 3/4 | 8/10 | 4/9 | 2/4 | 2/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/5 | 2/5 | 3/5 | 3/8 | 1/7 | 3/8 | 3/3 | 1/1 | 3/4 | 5/10 | 8/9 | 2/4 | 5/6
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 5/5 | 5/5 | 8/8 | 7/7 | 8/8 | 3/3 | 1/1 | 4/4 | 10/10 | 9/9 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADCT-301 Monotherapy 20 µg/kg (N=3) | ADCT-301 Monotherapy 30 µg/kg (N=5) | ADCT-301 Monotherapy 45 µg/kg (N=5) | ADCT-301 Monotherapy 60 µg/kg (N=5) | ADCT-301 Monotherapy 80 µg/kg (N=8) | ADCT-301 Monotherapy 100 µg/kg (N=7) | ADCT-301 Monotherapy 125 µg/kg (N=8) | ADCT-301 Monotherapy 150 µg/kg (N=3) | ADCT-301 Combination Therapy 20 µg/kg + Pemb (N=1) | ADCT-301 Combination Therapy 30 µg/kg + Pemb (N=4) | ADCT Combination Therapy 45 µg/kg + Pemb (N=10) | ADCT Combination Therapy 60 µg/kg + Pemb (N=9) | ADCT Combination Therapy 80 µg/kg + Pemb (N=4) | ADCT Combination Therapy 100 µg/kg + Pemb (N=6)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Immune-mediated adverse reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADCT-301 Monotherapy 20 µg/kg (N=3) | ADCT-301 Monotherapy 30 µg/kg (N=5) | ADCT-301 Monotherapy 45 µg/kg (N=5) | ADCT-301 Monotherapy 60 µg/kg (N=5) | ADCT-301 Monotherapy 80 µg/kg (N=8) | ADCT-301 Monotherapy 100 µg/kg (N=7) | ADCT-301 Monotherapy 125 µg/kg (N=8) | ADCT-301 Monotherapy 150 µg/kg (N=3) | ADCT-301 Combination Therapy 20 µg/kg + Pemb (N=1) | ADCT-301 Combination Therapy 30 µg/kg + Pemb (N=4) | ADCT Combination Therapy 45 µg/kg + Pemb (N=10) | ADCT Combination Therapy 60 µg/kg + Pemb (N=9) | ADCT Combination Therapy 80 µg/kg + Pemb (N=4) | ADCT Combination Therapy 100 µg/kg + Pemb (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 3 (4) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 4 (4) | 2 (2) | 0 (0) | 4 (4) | 4 (5) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (3) | 1 (1) | 3 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 3 (3) | 0 (0) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (6) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (3) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 6 (6) | 7 (11) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Breakthrough pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 7 (9) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 5 (8) | 1 (1) | 3 (4)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT03621982/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT03621982/SAP_001.pdf